CLINICAL TRIAL: NCT06744855
Title: Effect of Semiconductor Embedded Therapeutic Gloves on the Mitigation of Hand Osteoarthritis: A Randomized, Double-Blinded, Placebo-Controlled Clinical Trial
Brief Title: Effect of Semiconductor Embedded Therapeutic Gloves for Hand Osteoarthritis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Altoona Center for Clinical Research (Network)
Collaborators: INCREDIWEAR HOLDINGS, INC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-24
Record Dates: First submitted 2024-11-05; First posted 2024-12-20 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Hand Osteoarthritis; Osteoarthritis
Keywords: Semiconductor embedded fabric gloves for Hand Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Semiconductor circulation gloves (Active Comparator): The gloves will have semiconductors embedded in the fabric.
  Interventions: Device: Non-invasive circulation gloves
- Placebo circulation gloves (Placebo Comparator): The gloves will look identical to the active circulation gloves, but will not have semiconductors embedded into the fabric
  Interventions: Device: Fabric gloves

INTERVENTIONS:
Device: Non-invasive circulation gloves — Non-invasive class I medical device, circulation gloves with semiconductors embedded in the fabric.
  Arms: Semiconductor circulation gloves
Device: Fabric gloves — These gloves will look and feel identical to the active circulation gloves, but will not have semiconductors embedded in the fabric.
  Arms: Placebo circulation gloves

SUMMARY:
The goal of this study is to evaluate change in symptoms using semiconductor embedded gloves for hand osteoarthritis.

DETAILED DESCRIPTION:
The semiconductor embedded fabric emits mid-level and far infrared waves and negative ions to the tissue which can increase circulation of both blood and lymph, plus facilitates the anti-inflammatory nitric oxide cascade by accelerating the binding of Calcium to Calmodulin. Nitric oxide down-regulates interleukin1 beta and inducible nitric oxide synthase in certain cell types, which leads to reduced cyclooxygenase-2 and prostaglandins-molecules responsible for causing inflammation and pain. Unlike other systemic COX-2 inhibitors such as nonsteroidal anti-inflammatory drugs (NSAIDs), targeted infrared and negative ion therapy stimulate localized reaction pathways, thereby reducing pain and inflammation. This study seeks to identify patient reported subjective and clinically measured objective outcomes for hand osteoarthritis pain management and hand function with application of semiconductor embedded fabric in the affected area.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with erosive hand OA, non-erosive hand OA, or first carpometacarpal joint OA with a Kellgren- Lawrence grade >1 as determined by radiographic assessments and the American College of Rheumatology (ACR) classification
2. Patients age 40-75
3. Patients who are willing and able to adhere to follow-up schedule and protocol guidelines.
4. Patients who are willing and able to sign corresponding research subject consent form.

Exclusion Criteria:

1. Patient has a history of neurological conditions, including multiple sclerosis or Parkinson's disease
2. Patient has had prior surgical treatment of the hands in the last 5 years or injection treatment in the last 6 months
3. Patient has secondary OA including causes such as gout, rheumatoid arthritis, psoriatic arthritis
4. Patient has used topical creams or gels for arthritic pain including nonsteroidal anti-inflammatory drugs, capsaicin, lidocaine, or counterirritants in the last 1 week
5. Patient has a history of carpal tunnel syndrome, cubital tunnel syndrome, or radial tunnel syndrome
6. Patient has a history of peripheral neuropathy
7. Patient has chronic pain conditions unrelated to hand condition
8. Patient has auto-immune or auto-inflammatory diseases
9. Patient has used tobacco within the last 90 days
10. Patient is not within the ages of 40-75
11. Patient has an active infection (local or systemic)
12. Patient is unwilling or unable to sign the corresponding research subject consent form
13. Patient meets any other criteria or has any other condition that, in the opinion of the investigator, would prevent them from completing the study or that, in the opinion of the investigator, would confound study results.

    -

    Exclusion Criteria:

    -

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain as measured by the Visual Analog Scale (VAS) | Baseline and weekly for 9 months
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. The minimum number is zero meaning no pain and maximum number is 10 meaning the most pain the patient has every felt in their entire life. Lower scores are ideal while higher scores are indicative of the patient in a lot of pain.

SECONDARY OUTCOMES:
Change in patient hand function as determined by the Australian Canadian Osteoarthritis Hand Index (AUSCAN) | Baseline, 3 months, 6 months, and 9 months
  The Australian/Canadian Osteoarthritis Hand Index (AUSCAN) is a self-administered questionnaire that assesses hand pain, stiffness, and function in patients with osteoarthritis. It is on a 5-point Likert scale, with pain severity questions and answer ranges from strongly disagree to strongly agree.
Change in patient hand function as determined by the Functional Index for Hand Osteoarthritis (FIHOA) | Baseline, 3 months, 6 months, and 9 months
  The Functional Index for Hand Osteoarthritis (FIHOA) is a self-administered patient specific questionnaire to assess the patient's function with hand osteoarthritis. It has 10 questions and is on a 4-point Likert scale with 0 = possible without difficulty • 1 = possible with slight difficulty • 2 = possible with important difficulty • 3 = impossible.
Change in patient grip strength | Baseline, 3 months, 6 months, and 9 months
  Patient's grip strength will be assessed with a hand dynamometer. The patient will squeeze the device with the patient's elbow at 90 degrees of flexion and wrist in 30 degrees of extension. A force output value in pounds (lbs) will be displayed and a higher number of force output indicates a stronger grip strength.
Radiographic changes as determined by hand x-rays. | Baseline and 9 months
  Change of the arthritic hand joint health such as reduction in osteophyte formation, presence of erosions, and joint space narrowing as measured by radiographic assessments compared to pre-treatment scans. The PI will determine if the arthritic hand has improved, stabilized, or worsened during the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Altoona Center for Clinical Research, Duncansville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Pre-approval to share data and data results must be obtained by the corporation.

REFERENCES:
- [Result] Marino K, Lee R, Lee P. Effect of Germanium-Embedded Knee Sleeve on Osteoarthritis of the Knee. Orthop J Sports Med. 2019 Oct 25;7(10):2325967119879124. doi: 10.1177/2325967119879124. eCollection 2019 Oct. PMID 31696136